CLINICAL TRIAL: NCT02991482
Title: A Multicentre Randomised Phase III Trial Comparing Pembrolizumab Versus Standard Chemotherapy for Advanced Pre-treated Malignant Pleural Mesothelioma
Brief Title: PembROlizuMab Immunotherapy Versus Standard Chemotherapy for Advanced prE-treated Malignant Pleural Mesothelioma
Acronym: PROMISE-meso
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Merck Sharp & Dohme LLC (Industry); Frontier Science Foundation, Hellas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 9-15; 2016-002062-31 (EudraCT Number); 3475-594 (Other: Merck Sharp Dohme)
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Results first posted 2022-02-07 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Pleural Mesothelioma Malignant Advanced
Keywords: MPM
MeSH Terms: interventions — pembrolizumab; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab arm (Experimental): Pembrolizumab is administrated at 200 mg fixed dose i.v. on day 1 of every 3 week cycle for a maximum or 2 years (expected maximum of 36 doses), or until progression of disease determined according to RECIST 1.1 criteria or lack of tolerability, or until the patient declines further treatment.
  Interventions: Drug: Pembrolizumab
- Standard chemotherapy arm (Active Comparator): Gemcitabine (i.v. 1000 mg/m2) or vinorelbine (i.v. 30 mg/m2, or p.o 60/80 mg/m2) chemotherapy will be chosen on a per patient basis and delivered according to local standards. Chemotherapy will be administered on days 1 and 8 of every 3-week cycle. A maximum number of treatment cycles is not mandated.
  Patients randomised to the control arm will be allowed to cross over to receive pembrolizumab at progression, if cross-over criteria are met. Pembrolizumab administration will follow the same schedule as for patients in the experimental arm, i.e. 200 mg fixed dose i.v. on day 1 of every 3-week cycle for a maximum of 2 years or until trial termination.
  Interventions: Drug: Gemcitabine; Drug: Vinorelbine

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab (MK-3475) is a potent and highly selective humanised monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. This blockade enhances functional activity of the target lymphocytes to facilitate tumour regression and ultimately immune rejection.
  Other Names: KEYTRUDA; MK-3475; SCH 900475
  Arms: Pembrolizumab arm
Drug: Gemcitabine — Gemcitabine replaces one of the building blocks of nucleic acids, in this case cytidine, during DNA replication. The process arrests tumour growth, as new nucleosides cannot be attached to the "faulty" nucleoside, resulting in apoptosis (cellular "suicide").
  Other Names: Gemzar
  Arms: Standard chemotherapy arm
Drug: Vinorelbine — Vinorelbine is a vinca alkaloid cytotoxic chemotherapy that is available in intravenous and oral preparations with EMA licenses in lung cancer and breast cancer. Vinorelbine blocks mitosis in phase G2-M, causing cell death in interphase or at the following mitosis.
  Other Names: Navelbine
  Arms: Standard chemotherapy arm

SUMMARY:
Trial comparing standard treatment (chemotherapy) with pembrolizumab treatment in patients with advanced pretreated malignant mesothelioma.

DETAILED DESCRIPTION:
Mesothelioma is an aggressive malignancy usually affecting the surfaces of body coelomic cavities. It most commonly originates from the pleura with a propensity to the lower parietal pleura and costo-diaphragmatic recess, and is almost always caused by asbestos exposure, with a usual lag time of 30 years between exposure and presentation. Outcomes for most patients are invariably fatal, with median survival from presentation around 9-12 months in most series due to difficulties in achieving a complete microscopic surgical resection and tumour relative chemo-refractoriness. Whilst initially considered rare, due to the demand of asbestos of all varieties associated with industrialization following the Second World War, the background incidence of mesothelioma of 1/million has risen to 40/million in some countries. In the UK, where substantial asbestos exposure continued until the 1970s, the death rate is the highest in the world with a current epidemic of new cases, predicted to continue for another 5-10 years. Two main histological subtypes of mesothelioma are identified. The epitheliod subtype is the commonest, accounting for around 40% of cases, whilst the sarcomatoid subtype is observed in 20% of cases; the latter being typically aggressive and chemorefractory. Around 35% cases have features of both epitheliod and sarcomatoid subtypes and are termed biphasic subtype.

For patients with pleural mesothelioma, in whom surgery is not considered appropriate, systemic chemotherapy (platinum combined with pemetrexed) remains the international standard of care. Cisplatin/pemetrexed is associated with a response rate of 41% and confers an OS advantage of 3 months over cisplatin alone, and is the only licensed systemic therapy for mesothelioma in Europe. Despite this, the median survival is 9-12 months from most series in unresectable cases. At relapse, after platinum-based chemotherapy, no anti-cancer systemic therapies are licensed. Whilst several small phase II studies and retrospective series have suggested potential efficacy for chemotherapy with agents including carboplatin/gemcitabine, or vinorelbine, none thus far have demonstrated efficacy benefit in a randomised study, with median PFS rates reported of about 3 months for both gemcitabine and vinorelbine. There is therefore a huge unmet need for effective therapy for patients with relapsed pleural mesothelioma. The largest trial ever performed of systemic therapy in relapsed pleural mesothelioma in 661 patients documented the natural outcome of this group of relapsed mesothelioma patients, reporting a median OS of 27.1 weeks (6 months) and median PFS for 6.1 weeks (1.5 months) for placebo.

Programmed cell death-1 (PD-1) is a co-inhibitory molecule at the immunological synapse that acts as a major regulator of adaptive immunity, and is exploited by tumour cells to result in adaptive immune resistance (tolerance). This occurs when PD-1 binds to the ligands PD-L1 (B7H1) or PD-L2, which are expressed on many tumour types. High PD-L1 expression on tumours is associated with poorer outcomes. Mesothelioma has been shown to express PD-L1, with a small study identifying PDL1 expression in up to 40% of mesotheliomas. Moreover, immunologically-mediated inflammation is known to be a key driver for mesothelioma development via the Nalp3 imflammasome.

Pembrolizumab (MK-3475) is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.

There is a need to identify new ways for the systemic therapy of malignant mesothelioma and immune checkpoint inhibition is a promising way forward. Results from the proposed trial will contribute to overcoming tumour-specific immune suppression with immune checkpoint inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant pleural mesothelioma (all subtypes are eligible)
* Progressing after or on previous platinum based chemotherapy.
* Availability of tumour tissue for translational research.
* Female and male patients aged 18 years or over.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Life expectancy of at least 3 months.
* Measurable or evaluable disease according to RECIST 1.1 criteria.
* Adequate renal function
* Creatinine 1.5 × Upper Limit of Normal (ULN) OR Calculated creatinine clearance 40 mL/min (using the Cockroft-Gault formula).
* Adequate haematological function
* Haemoglobin 90 g/L or 5.6 mmol/L
* White Blood Cell (WBC) 1.0 × 109/L
* Lymphocytes 0.5 g/L
* Absolute neutrophils count (ANC) 1.5 × 109/L
* Platelet count 100 × 109/L.
* Adequate liver function
* ALT and AST 2.5 × ULN. If the patient has liver metastases, ALT and AST must be ≤5 × ULN.
* Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must have a negative serum or urine pregnancy test within 35 days before randomisation (the test has to be repeated 72 hours before pembrolizumab treatment start).
* Written informed consent must be signed and dated by the patient and the investigator prior to any trial-related intervention including the submission of mandatory biomaterial.

Exclusion Criteria:

* Prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), anti-programmed cell death ligand 2 (anti-PD-L2), anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Prior therapy with gemcitabine or vinorelbine.
* Known active central nervous system metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to randomisation and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to randomisation. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Known or suspected hypersensitivity to pembrolizumab or any of its excipients.
* Known unstable or unresolved surgical or chemotherapy-related toxicity that would compromise the patient's capacity to participate in the trial.
* Previous allogeneic tissue/solid organ transplant.
* Live vaccines within 30 days prior to first dose of pembrolizumab.
* Regular intake of immune-modulating drugs (such as interferon, methotrexate).
* History of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (i.e. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) or topical therapy (e.g., steroids) for psoriasis or eczema is not considered a form of systemic treatment.
* Ongoing clinically serious infections requiring systemic antibiotic or antiviral, antimicrobial, or antifungal therapy.
* Human immunodeficiency virus (HIV) infection.
* Known active hepatitis B or hepatitis C.
* Known history of active tuberculosis.
* Patients with diagnosed immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to randomisation.
* Patients with other serious diseases or clinical conditions, including but not limited to uncontrolled active infection and any other serious underlying medical condition that could affect the patient's capacity to participate in the trial.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the trial or evaluation of the trial results.
* Women who are pregnant or in the period of lactation.
* Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the trial and up to 120 days following cessation of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Popat, MD, Study Chair — Royal Marsden NHS Foundation Trust; Alessandra Curioni-Fontecedro, MD, Study Chair — University Hospital, Zürich
Locations (15):
- Spain (3):
  - Hospital Teresa Herrera, A Coruña
  - ICO Hospitalet, Barcelona
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Switzerland (5):
  - Kantonsspital Aarau, Aarau
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital Winterthur, Winterthur
  - University Hospital Zürich, Zurich
- United Kingdom (7):
  - Maidstone and Tunbridge Wells NHS Trust, Kent Oncology Centre, Maidstone, Kent
  - Addenbrooke's Hospital, Cambridge
  - Clatterbridge Cancer Centre, Liverpool
  - Royal Marsden Hospital, London
  - Guy's and St Thomas' Hospital, London
  - Plymouth Hospitals NHS Trust, Plymouth
  - Weston Park Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herbst RS, Baas P, Kim DW, Felip E, Perez-Gracia JL, Han JY, Molina J, Kim JH, Arvis CD, Ahn MJ, Majem M, Fidler MJ, de Castro G Jr, Garrido M, Lubiniecki GM, Shentu Y, Im E, Dolled-Filhart M, Garon EB. Pembrolizumab versus docetaxel for previously treated, PD-L1-positive, advanced non-small-cell lung cancer (KEYNOTE-010): a randomised controlled trial. Lancet. 2016 Apr 9;387(10027):1540-1550. doi: 10.1016/S0140-6736(15)01281-7. Epub 2015 Dec 19. PMID 26712084
- [Background] Robinson BW, Musk AW, Lake RA. Malignant mesothelioma. Lancet. 2005 Jul 30-Aug 5;366(9483):397-408. doi: 10.1016/S0140-6736(05)67025-0. PMID 16054941
- [Background] Fennell DA, Gaudino G, O'Byrne KJ, Mutti L, van Meerbeeck J. Advances in the systemic therapy of malignant pleural mesothelioma. Nat Clin Pract Oncol. 2008 Mar;5(3):136-47. doi: 10.1038/ncponc1039. PMID 18227828
- [Background] Rake C, Gilham C, Hatch J, Darnton A, Hodgson J, Peto J. Occupational, domestic and environmental mesothelioma risks in the British population: a case-control study. Br J Cancer. 2009 Apr 7;100(7):1175-83. doi: 10.1038/sj.bjc.6604879. Epub 2009 Mar 3. PMID 19259084
- [Background] Tsiouris A, Walesby RK. Malignant pleural mesothelioma: current concepts in treatment. Nat Clin Pract Oncol. 2007 Jun;4(6):344-52. doi: 10.1038/ncponc0839. PMID 17534390
- [Background] Vogelzang NJ, Rusthoven JJ, Symanowski J, Denham C, Kaukel E, Ruffie P, Gatzemeier U, Boyer M, Emri S, Manegold C, Niyikiza C, Paoletti P. Phase III study of pemetrexed in combination with cisplatin versus cisplatin alone in patients with malignant pleural mesothelioma. J Clin Oncol. 2003 Jul 15;21(14):2636-44. doi: 10.1200/JCO.2003.11.136. PMID 12860938
- [Background] Krug LM, Kindler HL, Calvert H, Manegold C, Tsao AS, Fennell D, Ohman R, Plummer R, Eberhardt WE, Fukuoka K, Gaafar RM, Lafitte JJ, Hillerdal G, Chu Q, Buikhuisen WA, Lubiniecki GM, Sun X, Smith M, Baas P. Vorinostat in patients with advanced malignant pleural mesothelioma who have progressed on previous chemotherapy (VANTAGE-014): a phase 3, double-blind, randomised, placebo-controlled trial. Lancet Oncol. 2015 Apr;16(4):447-56. doi: 10.1016/S1470-2045(15)70056-2. Epub 2015 Mar 20. PMID 25800891

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Chemotherapy Arm: Gemcitabine (i.v. 1000 mg/m2) or vinorelbine (i.v. 30 mg/m2, or p.o 60/80 mg/m2) chemotherapy will be chosen on a per patient basis and delivered according to local standards. Chemotherapy will be administered on days 1 and 8 of every 3-week cycle. A maximum number of treatment cycles is not mandated.
  Patients randomised to the control arm will be allowed to cross over to receive pembrolizumab at progression, if cross-over criteria are met. Pembrolizumab administration will follow the same schedule as for patients in the experimental arm, i.e. 200 mg fixed dose i.v. on day 1 of every 3-week cycle for a maximum of 2 years or until trial termination.
  Gemcitabine: Gemcitabine replaces one of the building blocks of nucleic acids, in this case cytidine, during DNA replication. The process arrests tumour growth, as new nucleosides cannot be attached to the "faulty" nucleoside, resulting in apoptosis (cellular "suicide").
  Vinorelbine: Vinorelbine is a vinca alkaloid cytotoxic chemotherapy that is available in intravenous and oral preparations with EMA licenses in lung cancer and breast cancer. Vinorelbine blocks mitosis in phase G2-M, causing cell death in interphase or at the following mitosis.
Period: Overall Study
Arm/Group | Pembrolizumab Arm | Standard Chemotherapy Arm
Started | 73 | 71
Crossed-over to Pembrolizumab at Progression | 0 | 45
Completed | 8 | 5
Not Completed | 65 | 66
Not completed — Disease progression | 56 | 47
Not completed — Death | 4 | 4
Not completed — Adverse Event | 1 | 6
Not completed — Patient decision | 1 | 1
Not completed — Physician Decision | 0 | 6
Not completed — Clinical deterioration | 1 | 0
Not completed — Patient feeling too unwell | 1 | 0
Not completed — Worsening of performance status | 0 | 1
Not completed — Death prior to study drug initiation | 1 | 0
Not completed — Consent withdrawal prior to study drug initiation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab Arm | Standard Chemotherapy Arm | Total
Number analyzed (Participants) | 73 | 71 | 144
Age, Continuous [Median (Full Range); unit: years] | 69.0 [52.0 to 83.0] | 71.0 [53.0 to 83.0] | 70.0 [52.0 to 83.0]
Age, Customized [Count of Participants; unit: Participants]
  Age category: <70 years | 42 | 29 | 71
  Age category: ≥70 years | 31 | 42 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 58 | 60 | 118
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 54 | 53 | 107
  Switzerland | 13 | 14 | 27
  Spain | 6 | 4 | 10
Histologic subtype [Count of Participants; unit: Participants]
  Epithelioid | 66 | 62 | 128
  Non-epithelioid | 7 | 9 | 16
Smoking history [Count of Participants; unit: Participants]
  Current | 5 | 4 | 9
  Former (≥100 cigarettes in the past during the whole life) | 34 | 28 | 62
  Never (0-99 cigarettes during the whole life) | 33 | 39 | 72
  Unknown/Missing | 1 | 0 | 1
ECOG performance status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction; 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2: Ambulatory and capable of all selfcare but unable to carry out any work activities, up and about more than 50% of waking hours.
  Of note, although an ECOG performance status (PS) of 0 or 1 was mandatory to be included in the study, one patient was allowed to enter the study with ECOG PS of 2 due to leg braces.
  Participants
    0 | 21 | 14 | 35
    1 | 51 | 57 | 108
    2 | 1 | 0 | 1
EORTC score [Count of Participants; unit: Participants] — EORTC prognostic score (EPS) was calculated based on Fennell et al.(2005) prognostic model. This model takes into account WBC count, ECOG PS, histologic subtype and gender. A value of smaller or equal to 1.27 signifies a "good prognosis" while a value of more than 1.27 a "poor prognosis".
  Participants
    Good prognosis | 45 | 54 | 99
    Poor prognosis | 28 | 17 | 45
Prior treatment [Count of Participants; unit: Participants]
  Carboplatin/Pemetrexed | 27 | 27 | 54
  Cisplatin/Pemetrexed | 24 | 22 | 46
  Platinum+/-Pemetrexed+/-Other | 13 | 17 | 30
  Cisplatin/Pemetrexed and Carboplatin/Pemetrexed | 7 | 1 | 8
  Missing | 2 | 4 | 6
PD-L1 Tumour proportion score [Count of Participants; unit: Participants] — PD-L1 expression (PD-L1 tumor proportion score) was evaluated by immunohistochemistry (IHC) assay using clone SP263. PD-L1 was quantified as number of positive cells and scored as percentage of PD-L1 positive cells within tumor region. The following classification of PD-L1 scoring was used: 0 to <1% positive tumor cells; 1 to <20% positive tumor cells; >=20% positive tumor cells; Not Evaluable; Not scored.
  Participants
    <1% | 36 | 30 | 66
    1-20% | 20 | 18 | 38
    ≥20% | 11 | 14 | 25
    Not evaluable | 2 | 4 | 6
    Not scored | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Assessed by Independent Radiological Review
Description: To investigate whether treatment with pembrolizumab improves PFS, compared to standard, institutional choice chemotherapy, assessed according to RECIST 1.1 criteria based on independent radiological review; using Kaplan-Meier method and compared between the two treatment arms by a stratified log rank test.
Time Frame: Time from randomization of the first patient until database cutoff date for the primary PFS analysis (Sep 2017 - Feb 2019; approximately 1.5 years).
Population: All efficacy evaluations were conducted in the intent-to-treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab Arm | Standard Chemotherapy Arm
Number analyzed (Participants) | 73 | 71
months | 2.5 [2.1 to 4.2] | 3.4 [2.2 to 4.3]
Statistical Analysis 1: Comparison: Pembrolizumab Arm vs Standard Chemotherapy Arm; Test type: Superiority; p = 0.76, Log Rank

2. Secondary Outcome: Objective Response Rate by Independent Radiological Review
Description: Defined as the best overall response (complete or partial response) across all assessment time-points from randomisation to end of trial treatment, determined by RECIST 1.1 criteria.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab Arm | Standard Chemotherapy Arm
Number analyzed (Participants) | 73 | 71
percentage of participants | 21.9 [13.1 to 33.1] | 5.6 [1.6 to 13.8]

3. Secondary Outcome: Overall Survival.
Description: Defined as time from the date of randomisation until death from any cause. Censoring will occur at the last follow-up date.
Time Frame: Time from randomization of the first patient until database cutoff date for the OS analysis (Sep 2017 - Aug 2019; approximately 2 years).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab Arm | Standard Chemotherapy Arm
Number analyzed (Participants) | 73 | 71
months | 10.7 [7.6 to 15.0] | 12.4 [7.4 to 16.1]

4. Secondary Outcome: Time to Treatment Failure.
Description: Time from from randomisation to discontinuation of treatment for any reason, including progression of disease, treatment toxicity, refusal and death, by Kaplan Meier method. Censoring will occur at the last follow-up date.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab Arm | Standard Chemotherapy Arm
Number analyzed (Participants) | 73 | 71
months | 2.8 [2.1 to 4.2] | 2.3 [2.1 to 3.9]

5. Secondary Outcome: Percentage of Patients Experienced AEs/SAEs
Description: The safety and tolerability of pembrolizumab treatment will be assessed through analysis of the worst grade of toxicity/adverse events according to CTCAE v4.0 criteria observed over the whole treatment period. Adverse events are collected from study treatment initiation to 30 days after treatment is ceased for any reason. Serious adverse events and events of clinical interest are collected within 90 days after last dose of trial treatment.
Time Frame: as for outcome 1
Population: Safety evaluation was conducted in the as-treated (AT) population: all randomised patients that received at least one dose of trial treatment, with treatment assignments designed according to actual study treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Arm | Standard Chemotherapy Arm
Number analyzed (Participants) | 72 | 70
Participants
  Experienced any adverse event | 70 | 65
  Experienced treatment related adverse event | 50 | 52
  Experienced treatment related adverse event of grade 3-5 | 14 | 18
  Experienced treatment related adverse event leading to death | 1 | 1
  Experienced treatment related adverse event leading to treatment discontinuation | 5 | 5

6. Secondary Outcome: Progression Free Survival (PFS) Assessed by Investigator
Description: Investigator assessed PFS, from the date of randomisation until documented progression or death, if progression is not documented. Censoring occurs at the last tumor assessment.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab Arm | Standard Chemotherapy Arm
Number analyzed (Participants) | 73 | 71
months | 3.5 [2.1 to 4.2] | 3.7 [2.2 to 4.3]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from randomization of the first patient until database cutoff date for the primary PFS analysis (Sep 2017 - Feb 2019; approximately 1.5 years). All-Cause Mortality was assessed from the date of randomization up to 2 years. All-Cause Mortality was assessed from the date of randomization until database cutoff date for the OS analysis (Sep 2017 - Aug 2019; approximately 2 years).
Description: In the 'All Cause Mortality' section, number of at risk patients includes all randomized patients, while in the 'Serious Adverse Events' and 'Other (Not Including Serious) Adverse Events' sections, at risk patients refer to the population who received at least one dose of trial treatment (safety cohort).
Arm/Group | Pembrolizumab Arm | Standard Chemotherapy Arm
All-Cause Mortality (participants affected / at risk) | 48/73 | 44/71
Serious Adverse Events (participants affected / at risk) | 25/72 | 20/70
Other Adverse Events (participants affected / at risk) | 70/72 | 65/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab Arm (N=72) | Standard Chemotherapy Arm (N=70)
Lung infection (Infections and infestations) | 4 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Bronchial infection (Infections and infestations) | 2 | 1
Pain (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 1
Confusion (Psychiatric disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Hypophysitis (Immune system disorders) | 1 | 0
Infection NOS (Infections and infestations) | 0 | 1
Lower respiratory infection (Infections and infestations) | 1 | 0
Non-neutropaenic infection (Infections and infestations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab Arm (N=72) | Standard Chemotherapy Arm (N=70)
Fatigue (General disorders) | 28 | 32
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 20 | 10
Pain (General disorders) | 19 | 19
Constipation (Gastrointestinal disorders) | 17 | 23
Nausea (Gastrointestinal disorders) | 16 | 24
Diarrhea (Gastrointestinal disorders) | 16 | 26
Anorexia (Metabolism and nutrition disorders) | 12 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 | 2
Vomiting (Gastrointestinal disorders) | 10 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 3
Insomnia (Psychiatric disorders) | 8 | 5
Lung infection (Infections and infestations) | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2
Edema limbs (General disorders) | 6 | 4
Mucositis oral (Gastrointestinal disorders) | 5 | 9
Urinary tract infection (Infections and infestations) | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Bronchial infection (Infections and infestations) | 4 | 2
Flu like symptoms (General disorders) | 5 | 2
GGT increased (Investigations) | 5 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Weight loss (Investigations) | 5 | 3
Alanine aminotransferase increased (Investigations) | 4 | 4
Dry mouth (Gastrointestinal disorders) | 3 | 4
Headache (Nervous system disorders) | 4 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 2
Anemia (Blood and lymphatic system disorders) | 3 | 11
Neutrophil count decreased (Investigations) | 0 | 10
Abdominal pain (Gastrointestinal disorders) | 2 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 4
Fever (General disorders) | 2 | 5
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Depression (Psychiatric disorders) | 3 | 4
Paresthesia (Nervous system disorders) | 1 | 4
Oral thrush (Gastrointestinal disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/82/NCT02991482/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT02991482/SAP_001.pdf